CLINICAL TRIAL: NCT05280964
Title: Effect of a Novel Online Physician Group-Coaching Program to Reduce Burnout in Trainees: A Randomized Controlled Trial
Brief Title: Better Together: an Online Physician Coaching Program for Medical Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-2035
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Burnout; Self-compassion; Moral Injury; Impostor Phenomenon
Keywords: Burnout; Medical Education
MeSH Terms: conditions — Burnout, Psychological; Stress Disorders, Post-Traumatic; imposter syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Enrolled into a 6 month coaching program from January 1 2021 to June 30 2021
  Interventions: Behavioral: Better Together Physician Coaching
- Control/Wait-list (No Intervention): No intervention from January 1 2021 to July 1 2021 (they were offered the coaching program from July 1 2021-Dec 31 2021)

INTERVENTIONS:
Behavioral: Better Together Physician Coaching — 6 month, online group coaching program
  Arms: Intervention

SUMMARY:
This is a single-institution randomized controlled trial. 101 female residents were recurited from the University of Colorado School of Medicine. They enrolled beginning in January 2021 and participated in the coaching program for 6 months via a web-based system. Participants were randomized into either the intervention or wait-list control arm. Participants in the intervention arm began the 6-month coaching program in January, 2021. Participants in the wait-list control arm have received no additional resources from the Better Together program between January and June 2021. The wait-list control group was invited to begin the 6-month coaching program in July 2021. In December 2021, participants from both the intervention and wait-list control groups will be invited to complete a 2nd post survey (identical to the post-survey from June 2021). There will be no incentive for completion of the 2nd post survey. Finally, the longitudinal effect of the program will be assessed by offering the same survey measuring wellbeing via various indices to the intervention arm at 6 months (1/2022), 12 months (7/2022) and 18 months (1/2023) after their intervention. Participation in this survey will be completely voluntary and not incentivized/compensated.

DETAILED DESCRIPTION:
Background:

Positive psychology coaching programs demonstrate efficacy in reducing emotional exhaustion (a construct of burnout) and improving coping skills among residents but rely on substantial faculty development and coordination for participants. Considering the disproportionate burnout risk faced by women trainees in medicine, novel strategies to mitigate this risk is needed. Among a national sample of resident physicians, 60% screen positive for burnout. Compared to age-matched peers, residents are significantly more likely to experience burnout and have burnout persist into early careers. Female trainees are particularly vulnerable, with long-term consequences affecting professional development and success. Disproportionate burnout among women may be a contributor to the "leaky pipeline" in academic medicine, where women start their careers as 46% of the resident workforce yet represent only 25% of full professors and 18% of department chairs. Social connectedness and the practice of self-compassion are important intervention in reducing burnout and increasing resilience among residents. Positive psychology coaching programs have specifically had demonstrated efficacy in faculty and residents. Web-based group coaching programs have not been assessed for their potential to reduce burnout and improve resilience and well-being among trainees.

A. Outcome Measure(s):

1. participation (administrative data)
2. participant experience and reflection (interview)
3. measures of burnout and self-compassion as measured on a pre- and post- program survey including the Maslach Burnout Inventory (MBI) and Neff Self Compassion Score (SCS). Semi structured qualitative interviews will be led by a PRA upon completion of the 6-month pilot. The interview script will include questions about program content, participant experience, coping skills, interpersonal connectedness, personal and professional satisfaction, and general reflections.

Description of Population to be Enrolled:

This pilot study recruited individuals from the University of Colorado graduate medical education training programs. The pilot program is limited to female trainees who have greater than 1 year of training left in order to give trainees time to complete the program prior to graduation. Enrollment in the program is entirely voluntary and trainees can cease enrollment at any time.

Study Design and Research Methods:

This is a single-institution randomized controlled trial. 101 female residents were recruited from the University of Colorado School of Medicine. They enrolled beginning in January 2021 and participated in the coaching program for 6 months via a web-based system. The website is secure and only available for program participants. There are monthly modules with asynchronous, self-directed delivery, designed to mitigate the time constraints and faculty development required of traditional in-person coaching. Video recordings of group-coaching calls will be made available to the program participants via the secure website with the intent to allow participants to benefit from group coaching even if they aren't able to attend the calls live. These recordings do contain PHI of participants.

101 women trainees from 12 ACGME training programs enrolled in the program. Participants were randomized into either the intervention or wait-list control arm. Participants in the intervention arm began the 6-month coaching program in January, 2021. Participants in the wait-list control arm have received no additional resources from the Better Together program between January and June 2021.

All participants in both intervention and wait-list control groups will be invited to complete the quantitative post-program survey in June 2021. At the time of the post-program survey in 6/2021, the wait-list control group will not have received the coaching intervention. Following the quantitative and qualitative data collection, the control group was be offered the 6-month coaching program from July-December 2021.

The wait-list control group was invited to begin the 6-month coaching program in July 2021. In December 2021, participants from both the intervention and wait-list control groups will be invited to complete a 2nd post survey (identical to the post-survey from June 2021). There will be no incentive for completion of the 2nd post survey.

Finally, the longitudinal effect of the program will be assessed by offering the same survey measuring wellbeing via various indices to the intervention arm at 6 months (1/2022), 12 months (7/2022) and 18 months (1/2023) after their intervention. Participation in this survey will be completely voluntary and not incentivized/compensated.

ELIGIBILITY:
Inclusion Criteria:

* graduate medical education trainees (residents and fellows) at the University of Colorado
* Female identifying

Exclusion Criteria:

* Non trainees
* non- female identifying

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Trainees who identify as female, including transwomen, gender non-conforming, non-binary, and gender queer.
Enrollment: 101 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Burnout at 6 months, 12 months and 18 months | Baseline measurement, post-intervention measurements at 6 months, 12 months and 18 months
  The Maslach's burnout inventory is a 22-item measurement of worker burnout which assesses emotional exhaustion (EE), depersonalization (DP), and personal fulfillment (PF) domains. Possible scores range from 0-6 on a Likert scale for each item. Scores oof EE ≥ 27 points, DP ≥ 10, and PF <33 would indicate a high degree of burnout. Scores of EE≤18 points, DP≤5 points, and PF≥40 points would indicate a low degree of burnout.

SECONDARY OUTCOMES:
Change from baseline Self Compassion at 6 months, 12 months and 18 months | Baseline measurement, post-intervention measurements at 6 months, 12 months and 18 months
  Neff's Self-Compassion Scale - Short Form is a 12 item measurement of self-compassion with higher scores indicating improved or better levels of self compassion.
Change from baseline Imposter Syndrome at 6 months, 12 months and 18 months | Baseline measurement, post-intervention measurements at 6 months, 12 months and 18 months
  The Young Impostor Syndrome Scale is an 8 item measurement of imposter phenomenon with scores ≥ 5 indicating "yes" to presence of imposter phenomenon and scores less than 5 being negative for presence of imposter phenomenon.
Change from baseline Moral Injury at 6 months, 12 months and 18 months | Baseline measurement, post-intervention measurements at 6 months, 12 months and 18 months
  The Moral Injury Symptom Score for healthcare professionals is a 22 item measure of moral injury symptoms that assesses betrayal, guilt, shame, moral concerns, loss of trust, loss of meaning, difficulty forgiving, self-condemnation, religious struggle, and loss of religious/spiritual faith with scores of 60 or higher correlating with extreme problems, scores of 45-59 being moderate and scores of 30-45 being mild.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rotenstein LS, Torre M, Ramos MA, Rosales RC, Guille C, Sen S, Mata DA. Prevalence of Burnout Among Physicians: A Systematic Review. JAMA. 2018 Sep 18;320(11):1131-1150. doi: 10.1001/jama.2018.12777. PMID 30326495
- [Result] Pommier E, Neff KD, Toth-Kiraly I. The Development and Validation of the Compassion Scale. Assessment. 2020 Jan;27(1):21-39. doi: 10.1177/1073191119874108. Epub 2019 Sep 13. PMID 31516024
- [Result] Mantri S, Lawson JM, Wang Z, Koenig HG. Identifying Moral Injury in Healthcare Professionals: The Moral Injury Symptom Scale-HP. J Relig Health. 2020 Oct;59(5):2323-2340. doi: 10.1007/s10943-020-01065-w. PMID 32681398
- [Result] Villwock JA, Sobin LB, Koester LA, Harris TM. Impostor syndrome and burnout among American medical students: a pilot study. Int J Med Educ. 2016 Oct 31;7:364-369. doi: 10.5116/ijme.5801.eac4. PMID 27802178
- [Result] Dyrbye LN, Shanafelt TD, Gill PR, Satele DV, West CP. Effect of a Professional Coaching Intervention on the Well-being and Distress of Physicians: A Pilot Randomized Clinical Trial. JAMA Intern Med. 2019 Oct 1;179(10):1406-1414. doi: 10.1001/jamainternmed.2019.2425. PMID 31380892
- [Result] Palamara K, Chu JT, Chang Y, Yu L, Cosco D, Higgins S, Tulsky A, Mourad R, Singh S, Steinhauser K, Donelan K. Who Benefits Most? A Multisite Study of Coaching and Resident Well-being. J Gen Intern Med. 2022 Feb;37(3):539-547. doi: 10.1007/s11606-021-06903-5. Epub 2021 Jun 7. PMID 34100238
- [Derived] Mann A, Fainstad T, Shah P, Dieujuste N, Thurmon K, Dunbar K, Jones C. "We're all going through it": impact of an online group coaching program for medical trainees: a qualitative analysis. BMC Med Educ. 2022 Sep 13;22(1):675. doi: 10.1186/s12909-022-03729-5. PMID 36100880
- [Derived] Fainstad T, Mann A, Suresh K, Shah P, Dieujuste N, Thurmon K, Jones CD. Effect of a Novel Online Group-Coaching Program to Reduce Burnout in Female Resident Physicians: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2210752. doi: 10.1001/jamanetworkopen.2022.10752. PMID 35522281